CLINICAL TRIAL: NCT05841836
Title: A Prospective, Multi-center, Randomized Controlled, Non-inferiority Clinical Trial of the Safety and Efficacy of the Suture-Mediated Closure System for Percutaneous Closure of the Common Femoral Artery Puncture Site
Brief Title: The Safety and Efficacy of the Suture-Mediated Closure System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Zylox Medical Device Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zylox20220321
Record Dates: First submitted 2023-03-31; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Peripheral Arterial Disease; Arterial Puncture
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Suture-Mediated Closure System (Experimental): Produced by Zhejiang Zylox Medical Device Co., Ltd.
  Interventions: Device: the Suture-Mediated Closure System
- Perclose ProGlide Suture-Mediated Closure System (Active Comparator): Perclose® ProGlide Suture-Mediated Closure System
  Interventions: Device: Perclose ProGlide Suture-Mediated Closure System

INTERVENTIONS:
Device: the Suture-Mediated Closure System — To reduce the TTH(Time to hemostasis) and TTA(Time to ambulation)of common femoral artery(CFA) puncture site
  Arms: the Suture-Mediated Closure System
Device: Perclose ProGlide Suture-Mediated Closure System — To reduce the TTH(Time to hemostasis) and TTA(Time to ambulation)of common femoral artery(CFA) puncture site
  Arms: Perclose ProGlide Suture-Mediated Closure System

SUMMARY:
This was a prospective, multicenter, randomized, controlled, non-inferiority clinical study with the primary objective of validating the safety and efficacy of the Suture-Mediated Closure System for percutaneous closure of the common femoral artery puncture site.

DETAILED DESCRIPTION:
This study was a prospective, multicenter, randomized, controlled, non-inferiority clinical trial. It is planned to be conducted in multiple clinical trial institutions and enroll 228 subjects. Eligible subjects were randomly divided into the experimental group or the control group at a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 years old and 85 years old, randomized
* Patients who can be examined or treated with a common femoral artery puncture interventional catheter using a 5F to 22F sheath tube
* Patient(or their guardians) who submitted a written informed consent for the this trial

Exclusion Criteria:

* Known to be pregnant or lactating
* The diameter of femoral artery on the puncture side was less than 5mm
* Patients requiring anterograde puncture approach
* Have participated in or plan to participate in another clinical trial in the same period
* Known allergy to any components of the device, and/or contraindications to contrast agents and anticoagulants
* International normalized ratio (INR) >2.0
* Traumatic vascular injury at the approach site
* Systemic or local groin infection
* Cerebrovascular accident or myocardial infarction within 3 months
* An arterial catheter needs to be placed at the access site
* Morbidly obese (BMI ≥40 kg/m2)
* The entire common femoral artery wall assessed by ultrasound, calcification located in the anterior wall cut, the extent of more than 50% circumferential or common femoral artery stenosis ≥50
* Femoral artery aneurysm, arteriovenous fistula or pseudoaneurysm in common femoral artery
* Using a clip vessel occluder at the past ipsilateral femoral artery access site
* Use of a puncture point occlusion device at the ipsilateral femoral access site within the past 30 days
* Underwent an intervention via ipsilateral femoral artery puncture within the past 30 days or within the next 30 days
* Ipsilateral femoral vein sheath needed to be used
* Evidence of previous common femoral artery surgery on the same side (e.g., inguinal incision)
* Hematoma at ipsilateral arterial access
* Other circumstances that the investigator deemed inappropriate for participation in the trial.femoral artery aneurysm, arteriovenous fistula or pseudoaneurysm in common femoral artery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of major complications at the access site | 30 days after the procedure
  The number of subjects who experienced major complications as a proportion of the total number of subjects who used the vascular stapler system

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zhao, Master, Principal Investigator — First Affiliated Hospital of Chongqing Medical University; Hongfei Sang, M.D., Principal Investigator — Second Affiliated Hospital of Soochow University; Jianming Sun, M.D., Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Changsheng Shi, Master, Principal Investigator — The Third Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China